CLINICAL TRIAL: NCT07390695
Title: Gamified Exercise for Hardcore Smokers: A Quasi-Experimental Protocol for Improving Cardiorespiratory Fitness and Smoking Cessation
Brief Title: The Researchers Would Like to Conduct a Trial Using Gamified Exercise to Increase Cardiorespiratory Fitness and Intention to Quit Smoking Among Hardcore Smokers Who Are Also Physically Inactive.
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Gadjah Mada University (Other)
Responsible Party: Principal Investigator, Ahmad Hidayat, Principal Investigator, Gadjah Mada University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KE/FK/1453/EC/2024
Record Dates: First submitted 2025-12-04; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cardiorespiratory Fitness or Endurance; Smoking Cessation
Keywords: exercise; gamification; cardiorespiratory fitness; smoking cessation
MeSH Terms: conditions — Smoking Cessation; Motor Activity

STUDY DESIGN:
Intervention Model Description: One group quasi-experiment. Using one group that is involved in the whole stages of research (pre-test, intervention, post-test, and follow-up).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Gamification Team (Experimental): A group of 60 physically inactive hardcore smokers participated in this study using a gamified exercise within 12 12-week intervention.
  Interventions: Behavioral: Gamification of a structured exercise program

INTERVENTIONS:
Behavioral: Gamification of a structured exercise program — A structured exercise program with FITT-VP principles is gamified and delivered to 60 physically inactive hardcore smokers.

SUMMARY:
The goal of this quasi-experiment is to learn if a gamified exercise works to improve cardiorespiratory fitness in physically inactive hardcore smokers. It will also learn about the effects of smoking cessation. The main questions it aims to answer are:

* Does a gamification of a structured training program improve the cardiorespiratory fitness and smoking cessation behavior among smokers?
* Is there any mediating effect from the level of physical activity between a gamified exercise and cardiorespiratory fitness?
* Will the smokers engage in the gamified exercise within the 12-week intervention?

This is a no-control group. The quasi-experiment will be conducted within one group (paired data).

ELIGIBILITY:
Inclusion Criteria:

* hardcore smokers (min 20 cigarettes per day)
* being active smokers at least 1 year
* physically active (MET less than 600 MET minutes per week)

Exclusion Criteria:

* having any medical conditions that limit them to participation in a program training

Ages: 17 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — This study is only for male participants.
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Estimated Maximal Oxygen Uptake (VO2Max) Measured by the Cooper 12-Minute Run Test | Baseline (Week 0) and post-intervention (Week 13)
  Estimated cardiorespiratory fitness assessed using the Cooper 12-Minute Run Test. Participants are instructed to run or walk as far as possible within 12 minutes. The total distance covered (in meters) is used to estimate maximal oxygen uptake (VO2Max), expressed in milliliters per kilogram per minute (mL/kg/min). Higher VO2Max values indicate better cardiorespiratory fitness.

SECONDARY OUTCOMES:
Level of Physical Activity Measured by the World Health Organization Global Physical Activity Questionnaire (GPAQ) | Baseline (Week 0) and post-intervention (Week 13)
  Physical activity level assessed using the World Health Organization Global Physical Activity Questionnaire (GPAQ). The GPAQ measures physical activity across work, transport, and leisure domains. Total physical activity is calculated in metabolic equivalent task minutes per week (MET-minutes/week). Higher scores indicate higher levels of physical activity.
Intention to Quit Smoking Measured by the Intention to Quit Smoking Scale (IQSS) | Baseline (Week 0) and post-intervention (Week 13)
  Smoking cessation intention was assessed using the Intention to Quit Smoking Scale (IQSS) developed by Söyler and Yorulmaz (2024). The IQSS is a self-reported questionnaire consisting of multiple items rated on a Likert-type scale. Total scores range from 8 to 40, with higher scores indicating a stronger intention to quit smoking.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitas Gadjah Mada, Yogyakarta, Special Region of Yogyakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided